CLINICAL TRIAL: NCT00279591
Title: Near-Continuous, Noninvasive Blood Pressure Monitoring to Improve Outcomes in Pediatric Transport
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of technical support and supplies
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 48082; CUMG Grant
Record Dates: First submitted 2006-01-17; First posted 2006-01-19 (Estimated); Results first posted 2012-04-30 (Estimated); Last update posted 2012-04-30 (Estimated); Status verified 2012-04

CONDITIONS: Pediatric Patients With SIRS (Systemic Inflammatory Response Syndrome)
MeSH Terms: conditions — Systemic Inflammatory Response Syndrome

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Continuous Blood Pressure Monitoring (Active Comparator): Patients received continuous blood pressure monitoring the entire time they were in med flight to the hospital.
  Interventions: Device: Continuous blood pressure monitoring using (Dinamap) standard oscillometric blood pressure device
- Standard of care blood pressure monitoring (Placebo Comparator): Patients received the normal standard of care for blood pressure monitoring during the course of the med flight to the hospital.
  Interventions: Device: Standard of care blood pressure monitoring

INTERVENTIONS:
Device: Continuous blood pressure monitoring using (Dinamap) standard oscillometric blood pressure device — Continuous blood pressure monitoring of patients during med flight to hospital
  Arms: Continuous Blood Pressure Monitoring
Device: Standard of care blood pressure monitoring — Patients received the standard of care for blood pressure monitoring while en route to the hospital via med flight.
  Arms: Standard of care blood pressure monitoring

SUMMARY:
A randomized controlled trial compared the clinical outcomes of transported pediatric patients monitored with an oscillometric blood pressure device versus those monitored with a near-continuous, noninvasive blood pressure.

DETAILED DESCRIPTION:
94 transported patients were randomized to a control arm, monitored with a standard oscillometric blood pressure device (Dinamap), or an experimental arm, monitored with a near-continuous, noninvasive blood pressure device (Vasotrac).

ELIGIBILITY:
Inclusion Criteria:

1. Pediatric patients transported by Angel One to Arkansas Children's Hospital.
2. Age Group: 1 year - 17 years AND
3. Patients at risk of developing SIRS (Systemic Inflammatory Response Syndrome), according to the criteria below.

   i. The presence of at least two of the following four criteria (one of which must be abnormal temperature or leukocyte count): A. Core temperature of >38.5 C or <36 C. B. Tachycardia, defined as mean heart rate >95th percentile for age in absence of external stimulus, chronic drugs, or painful stimuli.

   C. Mean respiratory rate >95th percentile for age, or >10% immature neutrophils.

   OR
4. Patients with moderate or severe head trauma, at risk of developing secondary ischemic brain injury, according to the criteria below.

   i. Glasgow Coma scale <15 with one or more of the following: A. Mass lesion or cerebral edema on CT or MRI scan. B. Post-Traumatic Seizure. C. Multiple Trauma. D. Focal Neurologic Signs. E. Intubation for control of suspected intracranial hypertension.

   -

Exclusion Criteria:

1. Wrist circumference less than 11cm (minimum size for the Vasotrac device).
2. Contractures of the wrists, not allowing correct placement of the Vasotrac device.
3. Hematoma(s) located on both wrists from recent redial (<24hr) artery puncture.
4. Patients likely to proceed to brain death per assessment of the referring physician.
5. Patients being treated for malignant hypertension.

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 94 (Actual)
Dates: Start 2006-06; Primary Completion 2007-06 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Stroud, MD, Principal Investigator — University of Arkansas
Locations (1):
- Arkansas Children's Hospital, Little Rock, Arkansas, United States

REFERENCES:
- [Result] Stroud MH, Prodhan P, Moss M, Fiser R, Schexnayder S, Anand K. Enhanced monitoring improves pediatric transport outcomes: a randomized controlled trial. Pediatrics. 2011 Jan;127(1):42-8. doi: 10.1542/peds.2010-1336. Epub 2010 Dec 20. PMID 21173006

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Pediatric interfacility helicopter transport patients between May 2006 and June 2007.
Groups:
- Control Group: Oscillometric Blood Pressure Monitoring
- Intervention Group: Near Continuous Blood Pressure Monitoring
Period: Overall Study
Arm/Group | Control Group | Intervention Group
Started | 48 | 46
Completed | 48 | 46
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group | Intervention Group | Total
Number analyzed (Participants) | 48 | 46 | 94
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 48 | 46 | 94
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 8.5 (5.6) | 6.5 (4.6) | 7.5 (5.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 16 | 36
  Male | 28 | 30 | 58
Region of Enrollment [Number; unit: participants]
  United States | 48 | 46 | 94

OUTCOME MEASURES:

1. Primary Outcome: The Difference in Hospital Length of Stay Between Those Who Received Continuous Blood Pressure Monitoring and Those Who Received Standard of Care
Description: This is the total number of participants analyzed for the intervention group and the total number of participants analyzed for the control group and the total number of days that each group was analyzed overall.
Time Frame: Up to two weeks
Population: Intention to Treat
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 48 | 46
days | 10.0 (13.8) | 5.4 (4.6)

2. Secondary Outcome: Intensive Care Unit (ICU) Length of Stay
Time Frame: Up to two weeks
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 48 | 46
days | 3.7 (4.5) | 2.8 (4.8)

3. Secondary Outcome: Total Number of Organ Failure Days (Multiple Organ Dysfunction) in the Intensive Care Unit (ICU)for the Control Group and Total Number of Organ Failure Days for the Intervention Group. Multiple Organ Dysfunction is Defined as Multiple Organ Failure.
Description: Total number of organ failure days is for each group as a whole.
Time Frame: Up to two weeks
Population: ITT
Measure: Number; unit: Days
Units Other Than Participants: Days
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 46 | 48
Number analyzed (Days) | 206 | 202
Days | 18 | 32
Statistical Analysis 1: Comparison: Intervention Group vs Control Group; Test type: Superiority or Other; p = 0.03, Fisher Exact

4. Secondary Outcome: Mean Daily Score Using the Therapeutic Intervention Scoring System (TISS-28) Scale.
Description: The Therapeutic Intervention Scoring System (TISS-28) is an illness severity score for the ICU. The TISS score can range from zero up to 78. The higher the score is, the more severe the illness. The TISS-28 scale measures the severity of a patient's illness.
Time Frame: Up to two weeks
Population: This is the total number of participants analyzed for the intervention group and the control group and the total number of days analyzed overall for the intervention group and the control group.
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Days
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 46 | 48
Number analyzed (Days) | 206 | 202
units on a scale | 22.4 (10.1) | 23.9 (10.1)

5. Secondary Outcome: Amount of Intravenous Fluid Resuscitation
Time Frame: At start of inter-facility transport, then every 15 minutes until arrival.
Measure: Mean (Standard Deviation); unit: ml/kg
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 48 | 46
ml/kg | 19.8 (22.2) | 9.9 (9.9)

ADVERSE EVENTS:
Arm/Group | Control Group | Intervention Group
Serious Adverse Events (participants affected / at risk) | 0/48 | 0/46
Other Adverse Events (participants affected / at risk) | 0/48 | 0/46

LIMITATIONS AND CAVEATS:
Small Sample Size. Halted prior to projected enrollment secondary to lack of technical support and supplies for near continuous BP measuring device.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes